CLINICAL TRIAL: NCT02140086
Title: Buteyko Based Remedial Breathing Therapy With Children With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARCIM Institute Academic Research in Complementary and Integrative Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RBT_03; RBT_03
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-03

CONDITIONS: Asthma
Keywords: asthma; Buteyko; remedial breathing; children
MeSH Terms: conditions — Asthma

ARMS (2):
- Buteyko based Remedial Breathing Therapy (Experimental): Buteyko based Remedial Breathing Therapy
  Interventions: Behavioral: Buteyko based Remedial Breathing Therapy
- Waiting List (No Intervention): Training in the course of the study

INTERVENTIONS:
Behavioral: Buteyko based Remedial Breathing Therapy — Buteyko based remedial Breathing Therapy after Dr. Buteyko
  Arms: Buteyko based Remedial Breathing Therapy

SUMMARY:
A randomized, controlled trial to investigate the effects of a buteyko based remedial breathing therapy on children with asthma regarding to their symptoms, use of medication and lung function tests.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent of the parents
* age 6- 15 years
* information and consent of the consulting doctor
* levels of asthma therapy 1-3

Exclusion Criteria:

* participation in another study

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2014-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Reduction of Betamimetics (-30%) at 3- and/or 6-month follow up | asthmaspezific parameters are measured before and after intervention as well as 3- and 6- month follow up

SECONDARY OUTCOMES:
Asthma Control Questionnaire (ACQ) | parameters are measured before and after intervention as well as 3- and 6- month follow up
  Scores of the ACQ (Asthma Control Questionnaire)
Paediatric Asthma Quality of Life Questionnaire (PAQLQ) | parameters are measured before and after intervention as well as 3- and 6- month follow up
  Scores of PAQLQ (Paediatric Asthma Quality of Life Questionnaire)
ARCIM Questionnaire (AFB) | parameters are measured before and after intervention as well as 3- and 6- month follow up
  Scores of the AFB (ARCIM Questionnaire) regarding to asthma symptoms of the last 3 month (AFB is not validated)
Peak Flow | parameters are measured before and after intervention as well as 3- and 6- month follow up
NO-measurement nasal and oral | parameters are measured before and after intervention as well as 3- and 6- month follow up
Buteyko-Questionnaire | parameters are measured before and after intervention as well as 3- and 6- month follow up
parameters of spirometry | parameters are measured before and after intervention as well as 3- and 6- month follow up
Paediatric asthma caregiver´s quality of life questionnaire (PACQLQ) | parameters are measured before and after intervention as well as 3- and 6- month follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Filderklinik, Filderstadt, Baden-Wurttemberg, Germany